CLINICAL TRIAL: NCT03231046
Title: Modality Augmentation for Navigation: Intuitive Fusion With Optical Lightweight Device (US/CBCT)
Acronym: MANIFOLD II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Clear Guide Medical (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGM 18-002
Record Dates: First submitted 2016-07-12; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Hepatic Biopsy or Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CBCT-US Fusion Arm (Experimental): Clear Guide SCENERGY, CBCT-US
  Interventions: Device: CBCT-US Fusion Arm
- EM Fusion or No Fusion Arm (Active Comparator)
  Interventions: Procedure: Hepatic Biopsy or Ablation

INTERVENTIONS:
Device: CBCT-US Fusion Arm — Use of Clear Guide SCENERGY for CBCT-US fusion guidance
  Other Names: Clear Guide SCENERGY, CBCT-US
  Arms: CBCT-US Fusion Arm
Procedure: Hepatic Biopsy or Ablation — Standard of Care
  Arms: EM Fusion or No Fusion Arm

SUMMARY:
The objective of this research is to evaluate functional validation of the CBCT-US fusion for the Clear Guide SCENERGY system, as well as to evaluate benefits derived from system performance.

DETAILED DESCRIPTION:
Human subjects are proposed to validate the CBCT-US fusion aspects of the Clear Guide SCENERGY product. For these modalities, Clear Guide Medical will work with the subcontract PI to determine the appropriate clinical procedure to evaluate (1) functional validation of the fusion system and (2) benefits derived from system performance. The selected procedure must be a single-patient interaction (i.e., no follow-up visits). Clinical studies will require approval through the subcontract's IRB. The Clear Guide SCENERGY will be compared to standard clinical practice (either no fusion or an electromagnetic-based fusion system). Clear Guide Medical plans to determine sample size based upon statistical powering for a predetermined clinically-meaningful difference (delta). This delta has not been selected, because this depends on the procedure selected. The anticipated sample size is expected to be around 100 subjects (i.e., 50 per arm), per modality. Blinding will be used, where possible. Clinician-related endpoints cannot be blinded due to obvious equipment differences. Subjects will be placed into treatment group by random. Retention strategies are unnecessary, as there will not be any planned follow-up visits or activities.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing radiological, oncological, or urological intervention procedures
* Able to give written informed consent

Exclusion Criteria:

* Unable to give informed consent
* Vulnerable populations and children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Success of needle placement | Immediately following intervention (within 2 hours)
  Distance between needle tip and target

IPD SHARING:
Plan to Share IPD: No